CLINICAL TRIAL: NCT06360016
Title: Protocol of Self-Regulation in Early Learners: The Role of Recreational Programs
Acronym: Protocol-RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Principal Investigator, Ezgi Ertüzün, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Protocol-RAP
Record Dates: First submitted 2024-03-09; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Self Regulation; Impulsive; Attention Difficulties; Emotion Regulation
Keywords: self regulation; recreational activities; preschoolers
MeSH Terms: conditions — Self-Control; Impulsive Behavior; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: pre and post-test with the control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol-RP (Experimental): The sample size was determined using the G-Power 3.01 program (G*Power 3.1 Manual, 2017), based on a Type I error of 0.05, a power of 0.95, and an effect size of f=0.55. According to these calculations, the sample size was set to a minimum of 10 individuals. Since the study was a pre-test post-test control group design and to prevent the reduction of internal validity due to any data loss, it was decided that each group (experimental and control) should have 20 participants.
  The school that formed the experimental group had only one preschool class, comprising 21 students.
  Interventions: Behavioral: Recreation Activity Program
- Control (No Intervention): The control group's school also had one preschool class, with 19 students making up the control group.

INTERVENTIONS:
Behavioral: Recreation Activity Program — Students in the study group were subjected to a 24-session RAP, including entertaining games. This program was conducted by the first-name researcher, who had completed their undergraduate education in preschool education and was supported by the second and third-named researchers as assistant instructors. The 24-session program, which included rhythm, balance, and patience acquisition games, was planned according to a game theory model that primarily aimed to entertain children. The program, aimed at developing children's self-regulation skills based on fundamental reflections of the model, would consist of simple rule-based entertaining games. Before the program's application, researchers provided information about the research and program to the experimental group, and verbal consent was obtained.
  Arms: Protocol-RP

SUMMARY:
Protocol of Self Regulation in Early Learners: The Role of Recreational Activity Program (RAP) RAP, which included fun games and lasted 24 sessions, was applied to the students in the study group. Twenty-four sessions include games that help gain rhythm, balance, and patience. The program is planned according to the game theory model, which aims to have fun for children. The program, which aims to develop children's self-regulation skills based on the essential reflections of the model, will include fun games with simple rules. Before the program was implemented, the researchers informed the experimental group about the research and the program, and verbal consent was obtained from the participants.

DETAILED DESCRIPTION:
The study titled "Protocol of Self-Regulation in Early Learners: The Role of Recreational Programs" focuses on the influence of structured recreational activities on the development of self-regulation skills among preschool children. Self-regulation is a crucial ability, facilitating children's academic performance, social behaviors, and emotional well-being.

RAP, which included fun games and lasted 24 sessions, was applied to the students in the study group. Twenty-four sessions include games that help gain rhythm, balance, and patience. The program is planned according to the game theory model, which aims to have fun for children. The program, which aims to develop children's self-regulation skills based on the essential reflections of the model, will include fun games with simple rules. Before the program was implemented, the researchers informed the experimental group about the research and the program, and verbal consent was obtained from the participants.

ELIGIBILITY:
Inclusion Criteria: Attending at least 22 sessions -

Exclusion Criteria:

-

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Self-Regulation Assessment | Pre-post test (before implemention and up to 24 weeks)
  Preschool Self-Regulation Assessment: The 'Preschool Self-Regulation Assessment' scale measured the self-regulation skills of the children. Developed by Smith-Donald et al. (2007), this assessment tool allows for a performance-based evaluation. The Practitioner's Assessment Form within the scale provides the evaluator with the opportunity to assess the child's emotions, attention level, and behaviors based on the interaction between the practitioner and the child. The Practitioner's Assessment Form is a rubric-type rating scale scored from 0 to 3. The Turkish adaptation of the scale was carried out by Tanrıbuyurdu and Yıldız in 2012. The factor analysis performed within the scope of construct validity has determined that the scale has a two-factor structure: Attention/Impulse Control and Positive Emotion. The scale consists of 16 items, and the reliability coefficient (α) of the entire scale has been determined as .83.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Yalçın Kişi, Student, Study Chair — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)